CLINICAL TRIAL: NCT06355180
Title: Esketamine Versus Electroconvulsive Therapy for Suicidal Ideation in Depressive Episodes: a Multicenter Randomized Controlled Trial
Brief Title: Esketamine vs ECT for Acute Suicidality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Wuhu Fourth People's Hospital (Unknown); The Second People's Hospital of Dali Bai Autonomous Prefecture (Unknown); Inner Mongolia Autonomous Region Mental Health Center (Unknown); Beijing Chaoyang District Third Hospital (Unknown); Beijing Daxing District Xinkang Hospital (Unknown)
Responsible Party: Principal Investigator, Gang Wang, President of Beijing Anding Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shoudufazhan2024-1-2122
Record Dates: First submitted 2024-03-27; First posted 2024-04-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Mood Disorders; Suicidal Ideation; Depressive Episode
Keywords: Esketamine; Depressive Episode; Suicidal Ideation; Mood Disorders; Multicenter; Randomized Controlled Study; Electroconvulsive therapy
MeSH Terms: conditions — Mood Disorders; Suicidal Ideation | interventions — Esketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is not feasible to blind participants and caregivers due to the distinct nature of the interventions. Outcome assessors (independent evaluators responsible for primary and secondary outcomes, such as SI and depression severity scores) and data analysts (personnel conducting statistical analyses) will remain blinded to group assignments through the use of randomized, coded data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous esketamine (Experimental): The experimental group will receive six administrations of adjunctive intravenous esketamine over a two-week intervention period, followed by a 10-week observational follow-up phase.
  Interventions: Drug: Esketamine
- Electroconvulsive therapy (Active Comparator): The control group will receive six administrations of adjunctive ECT over a two-week intervention period, followed by a 10-week observational follow-up phase.
  Interventions: Device: Electroconvulsive therapy

INTERVENTIONS:
Drug: Esketamine — The experimental group will receive intravenous esketamine hydrochloride. Participants will be asked to fast for 8 hours prior to administration. On treatment days, esketamine will be administered at a dose of 0.2 mg/kg, diluted in 0.9% sodium chloride solution. The infusion rate will be controlled with an infusion pump or syringe pump to ensure a minimum administration duration of 40 minutes. Treatment will be administered three times per week (the recommended interval between sessions is 1 to 2 days, adjustable based on clinical judgment) for two consecutive weeks, totaling six sessions. For participants demonstrating intolerance to either the dose of 0.2 mg/kg or the six-session regimen, investigators could modify the treatment protocol based on efficacy and safety assessments.
  Arms: Intravenous esketamine
Device: Electroconvulsive therapy — The control group will receive ECT. Prior to each session, participants will undergo safety evaluations and concomitant medication adjustments. Following an 8-hour fast and bladder evacuation, other preoperative preparations include intravenous administration of anticholinergic agents, short-acting anesthetics, and muscle relaxants. Electrodes will be placed unilaterally on the non-dominant hemisphere, with the seizure threshold determined via titration. The treatment will be administered three times per week (the recommended interval between sessions is 1 to 2 days, adjustable based on clinical judgment) for two consecutive weeks (six sessions in total). The protocol permitted regimen modifications for participants unable to tolerate the full course, based on efficacy and safety assessments.
  Arms: Electroconvulsive therapy

SUMMARY:
This study is a multicenter, randomized, non-inferiority, parallel-group clinical trial designed to evaluate the efficacy and safety of esketamine compared with electroconvulsive therapy (ECT) in the treatment of suicidal ideation during depressive episodes in patients with mood disorders. Furthermore, it aims to investigate the potential mechanisms underlying the anti-suicidal effects of esketamine.

DETAILED DESCRIPTION:
Suicide is a major global public health concern, yet current treatments for suicidal ideation (SI) remain limited in efficacy. This study evaluates whether a two-week course of six administrations of adjunctive intravenous esketamine is non-inferior to electroconvulsive therapy (ECT) in reducing SI among adults experiencing depressive episodes of mood disorders. This multicenter, randomized, non-inferiority, parallel-group trial will enroll 340 adults diagnosed with mood disorders with clinically significant SI during a depressive episode. Participants will be randomized in a 1:1 ratio to receive either six administrations of adjunctive intravenous esketamine or ECT over a two-week intervention period, followed by a 10-week observational follow-up phase (the total study duration will be 12 weeks). The primary outcome is the rate of remission of SI, defined as a Scale for Suicidal Ideation (SSI) score of less than 4, at the end of the two-week intervention. Secondary outcomes include comparative evaluations of treatment efficacy on depressive symptoms, cognitive function, quality of life, and social functioning, as well as safety. Exploratory outcomes include the identification of biomarker and neurobiological mechanisms of treatment response through analyses of biological specimens (blood, urine, and feces), multimodal magnetic resonance imaging (MRI), and electroencephalographic (EEG) measures.

ELIGIBILITY:
Inclusion Criteria (all five criteria must be met for an individual to be included):

1. Outpatients or inpatients aged 18 to 65 years (inclusive);
2. Having a current diagnosis of MDD or depressive episode in bipolar I/II disorder, established using the Mini-International Neuropsychiatric Interview, version 7.0.2 (MINI 7.0.2) and according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria;
3. Having a total score of 6 or more on the SSI at screening;
4. Having at least primary school education and the ability to comprehend assessment scales;
5. Having provided written informed consent.

Exclusion Criteria (an individual will be excluded if any one of the following criteria is met):

1. Having a current or historical diagnosis of neurodevelopmental, neurocognitive, psychotic, or substance-related disorders according to the DSM-5 criteria;
2. Having active delusions or hallucinations;
3. Suffering from severe/unstable systemic illness (illness affecting the central nervous system, cardiovascular, respiratory, hepatic, renal, endocrine, or hematologic systems) and judged by the investigator as unsuitable for participation;
4. Being judged by the investigator as at risk for substance abuse or addiction;
5. Using reserpine currently;
6. Contraindications to general anesthesia;
7. Having a history of seizure disorders (except for uncomplicated childhood febrile seizures);
8. Having severe drug or food allergies or allergy to any component of the study medication;
9. Having a history of treatment non-response or severe adverse reactions to esketamine, ketamine, or ECT;
10. Having participated in any other clinical trials within the three months before the enrollment;
11. Being pregnant, breastfeeding, or planning to become pregnant (for female participants) or planning to father a child (for male participants) during the study or within 12 weeks after the last dose of medication;
12. Being judged by researchers as unsuitable for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Remission rate of suicidal ideation | Baseline, after the sixth treatments (week 2)
  The Scale for Suicide Ideation (SSI) is a 19-item clinician-administered scale assessing the severity of suicidal ideation. Each item is scored from 0 to 2, yielding a total score ranging from 0 to 38, with higher scores indicating greater suicidal intent.
  The primary outcome is the rate of remission of suicidal ideation following the 2-week intervention (after 6 treatments), with the remission of suicidal ideation defined as having an SSI score of less than 4 (which indicates the absence of clinically significant suicidal ideation).

SECONDARY OUTCOMES:
Remission rate of suicidal ideation | Baseline, after the first treatment, after the third treatment, at week 4, week 8, and week 12
  Compare the suicide ideation remission rates between the two groups after the first treatment, after the third treatment, at week 4, week 8, and week 12. Suicide remission rate is defined as an SSI score of less than 4.
Rates of sustained remission and recurrence of suicide ideation | Baseline, after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Sustained remission: Defined as having SSI scores of less than 4 in two consecutive assessments.
  Recurrence: Defined as the emergence of suicidal behavior, an SSI score of 6 or more, or other composite indicators, following two consecutive assessments with SSI scores of less than 4.
  Compare the sustained remission rates and recurrence rates of suicidal ideation between the two groups after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12.
Changes in SSI Scores | Baseline, after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Compare the changes in SSI scores at each visit compared to baseline.
Changes in Columbia-Suicide Severity Rating Scale (C-SSRS) Scores | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Compare the changes in C-SSRS scores at each visit compared to baseline.
Response rate of depressive symptoms | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Response of depressive symptoms is defined as a 50% or more reduction from baseline in the Montgomery-Åsberg Depression Rating Scale(MADRS) score. Compare the response rates of depressive symptoms between the two groups at each visit.
Remission rate of depressive symptoms | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Remission of depressive symptoms is defined as a MADRS score of less than 12. Compare the remission rates of depressive symptoms between the two groups at each visit.
Changes in Montgomery Asberg Depression Rating Scale (MADRS) Scores | Baseline, after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Compare the changes in MADRS scores at each visit compared to baseline.
Changes in Quick Inventory of Depressive Symptoms Self Report (QIDS-SR-16) Scores | Baseline, after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Compare the changes in QIDS-SR-16 scores at each visit compared to baseline.
Changes in Clinical Global Impressions (CGI) Scores | Baseline, after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Compare the changes in CGI scores at each visit compared to baseline.
Changes in Short Form 12 Health Survey (SF-12) Scores | Baseline, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Self-reported questionnaire. The Short Form 12 Health Survey (SF-12) is a condensed version of the SF-36 health survey, designed to measure health-related quality of life. It includes 12 questions covering physical and mental health domains. These questions generate two main scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), which are standardized to a mean of 50 and a standard deviation of 10 in the general population.
  Compare the changes in SF-12 scores at each visit compared to baseline.
Changes in Sheehan Disability Scale (SDS) Scores | Baseline, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Self-reported questionnaire. Scale Range: 0-30. Higher scores indicate greater functional impairment.
  Compare the changes in SDS scores at each visit compared to baseline.
Changes in Digital Span Test (DST) Scores | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Self-reported questionnaire. Scale Range: 0-22. Higher scores indicate better working memory and attention.
  Compare the changes in DST scores at each visit compared to baseline.
Changes in Digit Symbol Substitution Test (DSST) Scores | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Self-reported questionnaire. Scale Range: 0-90. Higher scores indicate better cognitive processing speed and attention.
  Compare the changes in DSST scores at each visit compared to baseline.
Changes in Perceived Deficit Questionnaire for Depression 5-item (PDQ-D-5) Scores | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Self-reported questionnaire. Scale Range: 0-20. Higher scores indicate a greater perceived cognitive deficit.
  Compare the changes in PDQ-D-5 scores at each visit compared to baseline.
Changes in Young Mania Rating Scale (YMRS) Scores | Baseline, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Clinician rated scales. Scale Range: 0-60. Higher scores indicate more severe manic symptoms.
  Compare the changes in YMRS scores at each visit compared to baseline.
Changes in Clinician Administered Dissociative States Scale (CADSS) Scores | Baseline, after the 1st, 2nd, 3rd, 4th, 5th, and 6th esketamine treatments
  Clinician rated scales. Scale Range: 0-92. Higher scores indicate more severe dissociative symptoms.
  Compare the changes in CADSS scores at each esketamine treatment compared to baseline.
Adverse event | Baseline, after the first treatment, after the third treatment, after the sixth treatment (week 2), at week 4, week 8, and week 12
  Compare the incidence of adverse events and serious adverse events between the two groups.
Changes in neuroimaging metrics | Baseline, after the sixth treatments (week 2)
  Explore changes in neuroimaging metrics after the sixth treatment compared to baseline.
Changes in Electroencephalogram (EEG) metrics | Baseline, after the first treatment, after the sixth treatments (week 2)
  Explore changes in EEG metrics after the first and sixth treatment compared to baseline.
Changes in biological indicators | Baseline, after the first treatment, after the sixth treatments (week 2)
  Biological samples (blood, urine, and feces) will be collected from a subset of participants at baseline, after the first treatment, and after the sixth treatment for multi-omics profiling, including genomic, transcriptomic, epigenomic, metabolomic, microbiome, immunological, proteomic, and pharmacogenomic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, MD, Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (6):
- China (6):
  - Wuhu Fourth People's Hospital, Wuhu, Anhui
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang District Third Hospital, Beijing
  - Beijing Daxing District Xinkang Hospital, Beijing
  - The Second People's Hospital of Dali Bai Autonomous Prefecture, Dali
  - Inner Mongolia Autonomous Region Mental Health Center, Hohhot

IPD SHARING:
Plan to Share IPD: No